CLINICAL TRIAL: NCT06562426
Title: Relationship Between Maternal Awareness About Vitamin D for Under- Five Years Children and Their Health Status Outcomes: Cross Sectional Study
Brief Title: Relationship Between Maternal Awareness About Vitamin D for Under- Five Years Children and Their Health Status Outcomes
Acronym: Vit-D
Status: Active, not recruiting | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Eman Badr, Principal Investigator, Alexandria University
Other Study IDs: MAVD
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Maternal Care Patterns; Child Nutrition Disorders; Vitamin D Deficiency
Keywords: Vitamin D; Maternal Awareness; under-five children; Health status outcomes
MeSH Terms: conditions — Child Nutrition Disorders; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Descriptive group on vitamin D awareness — 300 mothers of under-five children will be recruited in the descriptive study to assess their awareness about vitamin D and observe children for their health status outcome. Three tools will be used which are; sociodemographic characteristics of children and their mothers, Mothers' Awareness of Vitamin D Structured Interview Schedule, and Health Status Outcomes of Under- Five Years Children. Permission to conduct the study will be obtained from the administrative authorities of the settings after an explanation of the aim of the study. Each mother will be interviewed individually to obtain characteristics of mothers and their children, as well as knowledge and performance regarding Vitamin D. Each child will be observed for the manifestation of vitamin D deficiency and to measure their weight and height.

SUMMARY:
The observational study aims to identify the relationship between maternal awareness about vitamin D for under-five-year-old children and their health status outcomes. The research Question is :

Is there a relationship between maternal awareness about vitamin D for under-five years children and their health status outcomes? Mothers of children under five will be interviewed about their knowledge and practices regarding vitamin D and their children's health status. Each child will be observed for the manifestation of vitamin D deficiency and to measure their weight and height.

DETAILED DESCRIPTION:
The observational study aims to identify the relationship between maternal awareness about vitamin D for under-five-year-old children and their health status outcomes. The research Question is :

Is there a relationship between maternal awareness about vitamin D for under-five-year-old children and their health status outcomes? This study will be conducted in the Outpatient and Inpatient Departments of Smouha Children's University Hospital (SCUH) at Alexandria and Matrouh General Hospital and Specialized Children's Hospital at Matrouh City.

Mothers of children under five will be interviewed about their knowledge and practices regarding vitamin D and their children's health status. Each child will be observed for the manifestation of vitamin D deficiency and to measure their weight and height. Written informed consent for participation will be obtained from a under five years mothers after an explanation of the aim of the study, their voluntary participation, and the right to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* under-five years

Exclusion Criteria:

* any associated neurological and chronic disorders

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 300 mothers and their under-five years children will attend the out-patient clinics.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Mothers' knowledge about Vitamin D Structured Interview Schedule to identify the mothers' knowledge regarding vitamin D supplementation. | through study completion, an average of 1 year.
  It includes multiple questions about; the importance of vitamin D, different sources of vitamin D, the appropriate age for starting vitamin D supplementation, frequency of giving vitamin D, the proper dose of vitamin D, the method for exposing children to sun baths the food rich with vitamin D and the source of her knowledge about vitamin D.
  All items will be scored at one point for known, and zero for unknown or incorrect answers. Mothers' responses for all knowledge items will be summed up and converted into percentages. All items will be scored at one point for known, and zero for unknown or incorrect answers. Mothers' responses for all knowledge items will be summed up and converted into percentages.
  Mothers' awareness levels will be categorized as follows:
  * Satisfied awareness level for ≥50%
  * Unsatisfied awareness level <50%

SECONDARY OUTCOMES:
Mothers' Performance About Vitamin D Supplementation Structured Interview Schedule to identify the mothers' performance regarding vitamin D supplementation. | through study completion, an average of 1 year.
  It includes multiple questions about mothers' practices for giving vitamin D supplementation, exposing the child to sun and giving the child food rich in vitamin D . Responses will be scored as one point for correctly done and zero for not done. A total score of mother's performance will be summed up and converted into percentages. Mothers' performance level will be categorized as following:
  * Satisfied performance level for ≥50%
  * Unsatisfied performance level <50%
Manifestations of vitamin D deficiency assessment record. Each item will be scored with presence or absence. | through study completion, an average of 1 year.
  It includes delayed closure of fontanels, delayed sitting and walking, delayed teething, muscles cramping, bow leg, knock knee and bone fracture.
Child's physical growth assessment sheet. | through study completion, an average of 1 year.
  It includes weight/kg., length/ height/cm. and Body mass index/kg/m2.
Previous medical and surgical history sheet. | through study completion, an average of 1 year.
  It includes items as exposure to any disease (pneumonia,...), previous hospitalization, cause of hospitalization, duration and previous surgery. Each item will be scored with No and Yes.

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Arafa Badr, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amaya-Montoya M, Duarte-Montero D, Nieves-Barreto LD, Montano-Rodriguez A, Betancourt-Villamizar EC, Salazar-Ocampo MP, Mendivil CO. 100 YEARS OF VITAMIN D: Dietary intake and main food sources of vitamin D and calcium in Colombian urban adults. Endocr Connect. 2021 Dec 9;10(12):1584-1593. doi: 10.1530/EC-21-0341. PMID 34766920
- [Background] Crincoli V, Cazzolla AP, Di Comite M, Lo Muzio L, Ciavarella D, Dioguardi M, Bizzoca ME, Palmieri G, Fontana A, Giustino A, Di Cosola M, Vincenzo B, Lovero R, Di Serio F. Evaluation of Vitamin D (25OHD), Bone Alkaline Phosphatase (BALP), Serum Calcium, Serum Phosphorus, Ionized Calcium in Patients with Mandibular Third Molar Impaction. An Observational Study. Nutrients. 2021 Jun 4;13(6):1938. doi: 10.3390/nu13061938. PMID 34200107
- [Background] Chang SW, Lee HC. Vitamin D and health - The missing vitamin in humans. Pediatr Neonatol. 2019 Jun;60(3):237-244. doi: 10.1016/j.pedneo.2019.04.007. Epub 2019 Apr 17. PMID 31101452
- [Background] Dinlen N, Zenciroglu A, Beken S, Dursun A, Dilli D, Okumus N. Association of vitamin D deficiency with acute lower respiratory tract infections in newborns. J Matern Fetal Neonatal Med. 2016 Mar;29(6):928-32. doi: 10.3109/14767058.2015.1023710. Epub 2015 Mar 19. PMID 25786473
- [Background] Luan Z, Ma Y, Xin Y, Qian J, Wang H. Possible Molecular Mechanisms by which Vitamin D Prevents Inflammatory Bowel Disease and Colitis-associated Colorectal Cancer. Curr Med Chem. 2017;24(9):911-917. doi: 10.2174/0929867323666161202153028. PMID 27915990
- [Background] Midtbo LK, Nygaard LB, Markhus MW, Kjellevold M, Lie O, Dahl L, Kvestad I, Froyland L, Graff IE, Oyen J. Vitamin D status in preschool children and its relations to vitamin D sources and body mass index-Fish Intervention Studies-KIDS (FINS-KIDS). Nutrition. 2020 Feb;70:110595. doi: 10.1016/j.nut.2019.110595. Epub 2019 Sep 19. PMID 31739173
- [Background] Nimitphong H, Park E, Lee MJ. Vitamin D regulation of adipogenesis and adipose tissue functions. Nutr Res Pract. 2020 Dec;14(6):553-567. doi: 10.4162/nrp.2020.14.6.553. Epub 2020 Aug 5. PMID 33282119